CLINICAL TRIAL: NCT05826418
Title: Dietary Optimization of Microbiome Recovery Following Fecal Microbiota Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: rCDI
Record Dates: First submitted 2023-03-17; First posted 2023-04-24 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Clostridium Difficile Infection; Fecal Microbiota Transplant
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEND diet (Experimental): patients being treated with FMT
  Interventions: Dietary Supplement: MEND diet
- mNICE (modified NICE) diet (Active Comparator): patients being treated with FMT
  Interventions: Dietary Supplement: mNICE diet

INTERVENTIONS:
Dietary Supplement: MEND diet — Participants will be asked to adhere to their randomized MEND diet for 4 weeks and FMT. The FMT being offered is part of standard clinical care, as recommended by current practice guidelines. They will complete bi-weekly IBS symptom score questionnaires and stool samples collection from consent to week 4. Following the 4-week intervention period patients will not be asked to adhere to a study diet.
  Arms: MEND diet
Dietary Supplement: mNICE diet — Participants will be asked to adhere to their randomized mNICEdiet for 4 weeks and FMT. The FMT being offered is part of standard clinical care, as recommended by current practice guidelines. They will complete bi-weekly IBS symptom score questionnaires and stool samples collection from consent to week 4. Following the 4-week intervention period patients will not be asked to adhere to a study diet.
  Arms: mNICE (modified NICE) diet

SUMMARY:
Recurrent Clostridioides difficle infection (rCDI) is a very significant problem in its own right and current fecal microbiota transplant (FMT) -based therapeutics will benefit from their optimization for this indication. It is likely that appropriate nutritional support coupled with microbiota-based drugs will yield superior clinical outcomes. However, both diet and gut microbiome are very complex. This project, which is based on a wealth of FMT experience, both clinical and investigational, over the past decade along with the novel techniques developed to identify dietary patterns and food groups that explain the most variation in gut microbiome, offers an ideal platform for performing systematic research in nutritional support that promotes gut microbiota health. The purpose is to Generate preliminary data with regards to tolerability of the Microbiota enhancing and nourishing diet (MEND) and its effects on the fecal microbiota in rCDI patients following FMT with the goal of developing larger clinical trials aimed to optimize post-FMT dietary management.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Clinical plans to undergo FMT therapy for treatment of rCDI (≥ 2 CDI recurrences following the initial episode within 1 year without contraindications to the treatment)
* Ability to comply with study requirements
* Age at least 18 years old

Exclusion Criteria:

* Underlying IBD
* History of stomach surgery or bowel resection
* Anticipated antibiotic exposure during the study period
* Advanced liver disease
* Ongoing alcohol or drug abuse
* Pregnancy
* Any reason felt by the investigator to complicate the feasibility of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Participant acceptance of the diet | 4 weeks
  Diet acceptability questionnaire: Includes 7 questions each with minimum and maximum values (1 and 7) and higher scores mean better outcomes.
Participant compliance with study procedures | intervention to 4 weeks
  24-hr dietary recalls will be used to assure adherence with the study diet

SECONDARY OUTCOMES:
Bacterial diversity | 1 week
  Shannon diversity index
Bacterial diversity | 4 weeks
  Shannon diversity index
Bacterial diversity | 3 months
  Shannon diversity index
Similarity to donor bacterial composition | 1 week
  Using SourceTracker: which uses modeling based on 16S rDNA sequencing, is the measurement tool used to assess the measure
Similarity to donor bacterial composition | 4 weeks
  Using SourceTracker: which uses modeling based on 16S rDNA sequencing, is the measurement tool used to assess the measure
Similarity to donor bacterial composition | 3 months
  Using SourceTracker
Bacterial composition | 1 week
  Relative abundance of specific bacteria previously documented to be predictive of successful FMT outcomes with respect to CDI recurrence
Bacterial composition | 4 weeks
  Relative abundance of specific bacteria previously documented to be predictive of successful FMT outcomes with respect to CDI recurrence
Bacterial composition | 3 months
  Relative abundance of specific bacteria previously documented to be predictive of successful FMT outcomes with respect to CDI recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Khoruts, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States